CLINICAL TRIAL: NCT04785612
Title: A Phase 2a, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Immunogenicity and Efficacy of A Respiratory Syncytial Virus Vaccine (RSVpreF) in A Virus Challenge Model in Healthy Adults
Brief Title: Study of RSVpreF Vaccination and RSV Challenge in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hvivo (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVO-CS-005
Record Dates: First submitted 2021-02-12; First posted 2021-03-08 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blinded, placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSVPreF (Experimental): A single intramuscular injection at a dose of 120 mcg reconstituted with sterile water for an 0.5 mL injection volume
  Interventions: Biological: RSVPreF
- Placebo (Placebo Comparator): A single intramuscular injection of Placebo to match active vaccine
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RSVPreF — A single dose of 120 mcg RSVpreF for intramuscular injection
  Arms: RSVPreF
Other: Placebo — A single Placebo dose for intramuscular injection to match experimental vaccine
  Arms: Placebo

SUMMARY:
In this randomised, placebo-controlled, double-blind Phase 2a study, healthy male and female participants 18-50 years of age will be given an investigational RSV vaccine (RSVpreF) and challenged with RSV one month later. The purpose of this research study is to assess the safety, immunogenicity and efficacy of RSVpreF using a human viral challenge model.

DETAILED DESCRIPTION:
Respiratory Syncytial Virus (RSV) is a common virus that affects all human age groups and can cause a range of respiratory disease such as bronchitis and lower respiratory infections. These serious illnesses affect infants and adults who are older especially if they are over 65, have chronic heart or lung disease or have a weakened immune system. Vaccination against RSV has the potential to be a highly beneficial and effective approach to reduce RSV disease in older adults and pediatric populations, however there is no current vaccine approved for the prevention of RSV infections.

RSVpreF is being developed to prevent RSV-associated moderate to severe lower respiratory tract disease in adults 60 years of age and in infants by active immunization of pregnant women.

This study is an exploratory proof-of-concept to assess the safety, immunogenicity and efficacy of RSVpreF using a human challenge model. The RSV challenge model is developed to help understanding the RSV disease and assess new vaccines by testing them in participants deliberately infected with the virus.

In this study, approximately 62 (up to 72) participants will be vaccinated with the investigational RSVpreF to account for withdrawals between vaccination and challenge. Participants will be randomised 1:1 to receive RSVpreF or placebo.

The study will consist of a vaccination phase, quarantine phase and a follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the participant and the Investigator.
* Aged between 18 and 50 years.
* In good health with no history, or current evidence, of clinically significant medical conditions, and no clinically significant test abnormalities that will interfere with participant safety.
* A documented medical history prior to enrolment.
* The following criteria are applicable to female participants participating in the study.

  1. Females of childbearing potential must have a negative pregnancy test prior to enrolment.
  2. Females of non-childbearing potential:

  <!-- -->

  1. Post-menopausal females; defined as having a history of amenorrhea for >12 months with no alternative medical cause, and /or by FSH level >40mIU/mL, confirmed by laboratory.
  2. Documented status as being surgically sterile (e.g. tubal ligation, hysterectomy, bilateral salpingectomy and bilateral oophorectomy).
* The following criteria apply to female and male participants:

  1. Female participants of childbearing potential must use one form of highly effective contraception. Hormonal methods must be in place from at least 2 weeks prior to the first study visit. The contraception use must continue until 28 days after the date of viral challenge/last dosing with IMP (whichever occurs last).
  2. Male participants must agree to the contraceptive requirements below at entry to quarantine and continuing until 28 days after the date of Viral challenge / last dosing with IMP (whichever occurs last): a. Use a condom with a spermicide to prevent pregnancy in a female partner or to prevent exposure of any partner (male and female) to the IMP. b. Male sterilisation with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate (please note that the use of condom with spermicide will still be required to prevent partner exposure). This applies only to males participating in the study. c. In addition, for female partners of child bearing potential, that partner must use another form of contraception such as one of the highly effective methods mentioned above for female participants.

     In addition to the contraceptive requirements above, male participants must agree not to donate sperm following discharge from quarantine until 28 days after the date of Viral Challenge/last dosing with IMP (whichever occurs last).
  3. True abstinence - sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant.
* Sero-suitable to the challenge virus.

Exclusion Criteria:

* History of, or currently active, symptoms or signs suggestive of upper or lower respiratory tract infection within 4 weeks prior to the first study visit.
* a) Any history or evidence of any other clinically significant or currently active systemic comorbidities including psychiatric disorders (includes participants with a history of depression and/or anxiety).

  b) And/or other major disease that, in the opinion of the Investigator, may put the participant at undue risk, or interfere with a participant completing the study and necessary investigations (e.g autoimmune disease or immunodeficiency).
* Participants who have smoked ≥ 10 pack years at any time [10 pack years is equivalent to one pack of 20 cigarettes a day for 10 years].
* A total body weight ≤ 50 kg and Body Mass Index (BMI) ≤18 kg/m2 and ≥30kg/m2.
* Females who:

  1. Are breastfeeding, or
  2. Have been pregnant within 6 months prior to the study.
* History of anaphylaxis-and/or a history of severe allergic reaction or significant intolerance to any food or drug or vaccine, including hypersensitivity to any of the constituents of the study vaccine, as assessed by the PI.
* Venous access deemed inadequate for the phlebotomy and cannulation demands of the study.
* a) Any significant abnormality altering the anatomy of the nose in a substantial way b) Any clinically significant history of epistaxis (large nosebleeds) within the last 3 months c) Any nasal or sinus surgery within 3 months
* a) Evidence of vaccinations with licensed live attenuated vaccines within the 4 weeks prior to the planned date of viral challenge/first dosing with IMP (whichever occurs first). Evidence of vaccinations with licensed vaccines which are not live attenuated within the 2 weeks prior to the planned date of viral challenge/first dosing with IMP (whichever occurs first).

  b) Intention to receive any vaccination(s) before at least 28 days after the viral challenge (NB. No travel restrictions will apply after the Day 28 Follow-up visit).
* Receipt of blood or blood products, or loss (including blood donations) of 550 mL or more of blood during the 2 months prior to the planned date of viral challenge/first dosing with IMP (whichever occurs first) or planned during the 2 months after the viral challenge.
* a) Receipt of any investigational drug within 3 months prior to the planned date of viral challenge/first dosing with IMP (whichever occurs first).

  b) Previous vaccination with any licensed or investigational RSV vaccine before enrolment into the study. c) Receipt of three or more investigational drugs within the previous 12 months prior to the planned date of viral challenge/first dosing with IMP (whichever occurs first).

  d) Prior inoculation with a virus from the same virus-family as the challenge virus.

  e) Prior participation in another human viral challenge study with a respiratory virus in the preceding 3 months, taken from the date of viral challenge in the previous study to the date of expected viral challenge in this study.

  f) Receipt of treatment with immunosuppressive therapy.
* a) Confirmed positive test for drugs of abuse and cotinine on first study visit. One repeat test allowed at PI discretion.

  b) History or presence of alcohol addiction, or excessive use of alcohol
* A forced expiratory volume in 1 second (FEV1) < 80%.
* Positive human immunodeficiency virus (HIV), active hepatitis A (HAV), B (HBV), or C (HCV) test.
* Those employed or immediate relatives of those employed at hVIVO, Pfizer or any vendor.
* Any other finding that, in the opinion of the Investigator, deems the Participant unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Mann, Study Director — Hvivo; Golam Kabir, MD, Principal Investigator — Hvivo
Locations (1):
- Golam Kabir, London, United Kingdom

REFERENCES:
- [Derived] Schmoele-Thoma B, Zareba AM, Jiang Q, Maddur MS, Danaf R, Mann A, Eze K, Fok-Seang J, Kabir G, Catchpole A, Scott DA, Gurtman AC, Jansen KU, Gruber WC, Dormitzer PR, Swanson KA. Vaccine Efficacy in Adults in a Respiratory Syncytial Virus Challenge Study. N Engl J Med. 2022 Jun 23;386(25):2377-2386. doi: 10.1056/NEJMoa2116154. PMID 35731653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 participants were to be enrolled and vaccinated with the study vaccine, with 62 participants challenged with the study virus.
Pre-assignment Details: 70 participants were consented and vaccinated to ensure that 62 were able to then be challenged with RSV-A Memphis 37b accounting for dropouts between vaccination and challenge.
Period: Overall Study
Arm/Group | RSVPreF | Placebo
Started | 35 | 35
Completed | 31 | 31
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSVPreF | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (6.46) | 27.1 (6.78) | 26.5 (6.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 25 | 25 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 31 | 34 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Viral Load-time Curve (VL-AUC) of RSV
Description: The VL-AUC of RSV determined by qRT-PCR from nasal wash samples collected twice daily starting two days post-viral challenge (Day +2) up to discharge from quarantine.
Time Frame: Day 2 to Day 12
Population: The primary analysis used the ITT (Intent-to-Treat) Challenge Analysis Set which included all participants randomly assigned to study intervention and who took a dose of study vaccine/placebo and were given viral challenge.
Measure: Median (Inter-Quartile Range); unit: h*log10 PFU/mL
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
h*log10 PFU/mL | 0.00 [0.0 to 19.02] | 96.65 [0.0 to 675.32]

2. Primary Outcome: Number of Participants With RT-PCR Confirmed (Detected) Incidence of Symptomatic Infection
Description: RT-PCR-confirmed symptomatic RSV infection defined as:
  - Two detectable qRT-PCR reported on 2 or more consecutive days (any two detectable (≥LLOD) qRT-PCR measurements reported over 4 consecutive scheduled timepoints).
  and
  - Either one or more positive clinical symptoms from different categories in the symptom scoring system or one Grade 2 symptom from any category
Time Frame: Day 2 to Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 2 | 15

3. Primary Outcome: Sum Total Symptoms Diary Card Score (TSS)
Description: The sum total symptoms score is the sum of all scores from the first assessment on Day 1 to the first assessment on Day 12 (34 assessments). Symptom scores were collected three times daily starting one day post-viral challenge (Day +1) up to discharge from quarantine using a participant self-reportable 13-symptoms card. Clinical symptoms include runny nose, stuffy nose, sneezing, sore throat, earache, malaise/tiredness, headache, muscle or joint ache, chilliness/feverishness, cough, chest tightness, shortness of breath, and wheeze. Participants scored symptoms from 0 (no symptoms) - 3 (severe). Shortness of breath and wheeze had an additional scoring option of grade 4. For each assessment, an individual total symptom score was derived as the total of the scores given to the 13 symptoms on that symptom score card. Individual total symptom scores ranged from 0 (if all symptoms graded 0) to 41 (if all symptoms graded 3 and shortness of breath and wheeze graded 4).
Time Frame: Day 1 to Day 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: score on a scale
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
score on a scale | 2.1 (199.8) | 28.9 (120.2)

4. Secondary Outcome: Number of Participants With RT-PCR Confirmed (Quantifiable) Incidence of Symptomatic Infection
Description: RT-PCR confirmed RSV infection defined as
  * Two quantifiable PCR measures reported on 2 or more consecutive days (any two quantifiable (≥LLOQ) qRT-PCR measurements reported over 4 consecutive scheduled timepoints), and
  * Either one or more positive clinical symptoms from different categories in the symptom scoring system or one Grade 2 symptom from any category
Time Frame: Day 2 to Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 0 | 13

5. Secondary Outcome: Number of Participants With Culture Lab-confirmed Reduction of Symptomatic RSV Infection
Description: Culture lab-confirmed symptomatic RSV infection defined as:
  * One quantifiable viral culture and
  * Either one or more positive clinical symptoms from different categories in the symptom scoring system or one Grade 2 symptom from any category
Time Frame: Day 2 to Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 0 | 11

6. Secondary Outcome: Peak Viral Load of RSV by qRT-PCR
Description: Reduction in Peak viral load of RSV determined by quantifiable qRT-PCR from nasal samples collected twice daily starting two days post-viral challenge (Day +2) up to discharge from quarantine.
Time Frame: Day 2 to Day 12
Measure: Median (Inter-Quartile Range); unit: log 10 copies/mL
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
log 10 copies/mL | 0.00 [0.0 to 3.1080] | 4.2 [0.0 to 6.9990]

7. Secondary Outcome: Peak Viral Load of RSV by Viral Culture
Description: Peak viral load of RSV determined by quantifiable viral culture from nasal samples collected twice daily starting two days post-viral challenge (Day +2) up to discharge from quarantine.
Time Frame: Day 2 to Day 12
Measure: Mean (Standard Deviation); unit: log 10 PFU/mL
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
log 10 PFU/mL | 0.00 (0.00) | 1.921 (2.3837)

8. Secondary Outcome: Duration of Quantifiable qRT-PCR Measurements
Description: Duration (time in hours) of quantifiable qRT-PCR measurements from nasal samples collected twice daily starting two days post-viral challenge (Day +2) up to discharge from quarantine.
Time Frame: Day 2 to Day 12
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
hours | 18.0 [11.8 to 54.4] | 131.6 [72.1 to NA] — NA - the upper quartile was not estimable due to more than 25% of participants being censored, as they had not met the required criteria, at the end of their observation period.

9. Secondary Outcome: Duration of Quantitative Viral Culture Measurements
Description: Duration (time in hours) of quantitative viral culture measurements from nasal samples collected twice daily starting two days post-viral challenge (Day +2) up to discharge from quarantine.
Time Frame: Day 2 to Day 12
Population: Only infected subjects are included in the analysis, hence 0 for RSVPreF and 13 for Placebo
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 0 | 13
hours |  | 83.1 [60.2 to 95.8]

10. Secondary Outcome: VL-AUC Determined by Quantitative Viral Culture
Description: VL-AUC of RSV as determined by quantitative viral culture on nasal samples starting two days post-viral challenge (Day +2) up to discharge from quarantine
Time Frame: Day 2 to Day 12
Measure: Mean (Standard Deviation); unit: h*log10 PFU/mL
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
h*log10 PFU/mL | 0.00 (0.00) | 91.91 (127.883)

11. Secondary Outcome: Area Under the Curve Over Time of Total Clinical Symptoms (TSS-AUC)
Description: Data presented is hours * score. TSS-AUC (trapezium rule) as measured by graded symptom scoring system collected 3 times daily starting Day +1 up to Day 12am using a participant self-reportable 13-symptoms card, the max number of diary cards included in the AUC calculation is 34, the maximum time period is 264hrs.
  Clinical symptoms included runny nose, stuffy nose, sneezing, sore throat, earache, malaise/tiredness, headache, muscle or joint ache, chilliness/feverishness, cough, chest tightness, shortness of breath, and wheeze. Participants scored symptom from 0 (no symptoms) - 3(severe). Shortness of breath and wheeze had an additional scoring option of grade 4. Dairy card total symptom scores ranged from 0 (if all symptoms graded 0) to 41 (if all symptoms graded 3 and shortness of breath and wheeze graded 4).
  The range of TSS AUC scores are between 0 and 10,824 hours*score (maximum of 264x41).
Time Frame: Day 1 to Day 12
Measure: Mean (Standard Deviation); unit: hours * score on a scale
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
hours * score on a scale | 52.85 (105.250) | 230.76 (277.988)

12. Secondary Outcome: Peak Symptoms Diary Card Score
Description: Peak TSS for each participant is defined as the diary card total with the worst score (highest). The symptom scoring system was collected three times daily starting one day post-viral challenge (Day +1) up to discharge from quarantine using a participant self-reportable 13-symptoms card. Clinical symptoms include runny nose, stuffy nose, sneezing, sore throat, earache, malaise/tiredness, headache, muscle or joint ache, chilliness/feverishness, cough, chest tightness, shortness of breath, and wheeze. Participants scored symptoms from 0 (no symptoms) - 3 (severe). Shortness of breath and wheeze had an additional scoring option of grade 4. For each assessment, an individual total symptom score was derived as the total of the scores given to the 13 symptoms on that symptom score card. Individual total symptom scores ranged from 0 (if all symptoms graded 0) to 41 (if all symptoms graded 3 and shortness of breath and wheeze graded 4).
Time Frame: Day 1 to Day 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
score on a scale | 1.3 (1.79) | 4.1 (3.92)

13. Secondary Outcome: Peak Daily Symptom Score
Description: Peak daily symptom score was derived, for each day from Day 1 to Day 12, as the maximum of the 3 total symptoms scores on that day, providing 11 scores each. The symptoms were collected three times daily starting one day post-viral challenge (Day +1) up to discharge from quarantine using a participant self-reportable 13-symptoms card. Clinical symptoms include runny nose, stuffy nose, sneezing, sore throat, earache, malaise/tiredness, headache, muscle or joint ache, chilliness/feverishness, cough, chest tightness, shortness of breath, and wheeze. Participants scored symptoms from 0 (no symptoms) - 3 (severe). Shortness of breath and wheeze had an additional scoring option of grade 4. For each assessment, an individual total symptom score was derived as the total of the scores given to the 13 symptoms on that symptom score card. Individual total symptom scores ranged from 0 (if all symptoms graded 0) to 41 (if all symptoms graded 3 and shortness of breath and wheeze graded 4).
Time Frame: Day 1 to Day 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
score on a scale
  Day 1 | 0.6 (1.38) | 0.2 (0.56)
  Day 2 | 0.4 (0.76) | 0.3 (0.70)
  Day 3 | 0.3 (0.69) | 0.2 (0.50)
  Day 4 | 0.3 (0.73) | 1.1 (2.16)
  Day 5 | 0.5 (1.48) | 1.6 (2.78)
  Day 6 | 0.6 (1.12) | 2.2 (2.77)
  Day 7 | 0.4 (0.71) | 2.5 (3.04)
  Day 8 | 0.3 (0.58) | 2.5 (3.30)
  Day 9 | 0.3 (0.51) | 1.3 (1.59)
  Day 10 | 0.2 (0.55) | 0.7 (1.03)
  Day 11 | 0.2 (0.75) | 0.8 (1.51)
  Day 12 | 0.0 (0.18) | 0.5 (1.89)

14. Secondary Outcome: Percentage Number of Participants With Grade 2 or Higher Symptoms
Description: Number (%) of participants with Grade 2 or higher symptoms (on any occasion from Day 1 to Day 12)
Time Frame: Day 1 to Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 5 | 16

15. Secondary Outcome: Number of Participants With an Occurrence of at Least Two Positive Quantifiable qRT-PCR Measurements on 2 or More Consecutive Days
Description: The number of participants with at least two quantifiable positive (≥LLOQ) qRT-PCR nasal sample measurements across 4 consecutive visits
Time Frame: Day 2 to Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 4 | 16

16. Secondary Outcome: Number of Participants With an Occurrence of at Least Two Positive Detectable qRT-PCR Measurements on 2 or More Consecutive Days
Description: The proportion of participants with at least two positive detectable qRT-PCR nasal sample measurements across 4 consecutive visits
Time Frame: Day 2 to Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 10 | 23

17. Secondary Outcome: Number of Participants With an Occurrence of at Least One Positive Quantitative Cell Culture Measurements
Description: The proportion of participants with at least one quantifiable positive (≥LLOQ) nasal sample viral culture starting two days post-viral challenge (Day+2) up to discharge from quarantine. Viral culture is only done for samples where qRT-PCR is positive (detectable), when the qRT-PCR is negative the viral culture is assumed to be 0 for any endpoint derivations.
Time Frame: Day 2 to Day 12
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
Participants | 0 | 13

18. Secondary Outcome: Total Mucus Weight
Description: Total weight of mucus produced starting one day post-viral challenge (Day +1) up to discharge from quarantine.
  The mean sum of all mucus produced from Day 1 to Day 12 is reported in data table.
Time Frame: Day 1 to Day 12
Measure: Mean (Standard Deviation); unit: g
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
g | 6.367 (9.8246) | 29.135 (36.2811)

19. Secondary Outcome: Total Tissue Number
Description: Total number of tissues used by participants starting one day post-viral challenge (Day +1) up to discharge from quarantine.
Time Frame: Day 1 to Day 12
Measure: Mean (Standard Deviation); unit: Tissues
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 31 | 31
Tissues | 16.9 (22.35) | 41.7 (44.80)

20. Secondary Outcome: Number of Solicited Local Reactions Within 7 Days After Vaccination
Description: Local reactions include pain at injection site, redness and swelling
Time Frame: 7 days post vaccination
Population: The number of participants who completed the vaccination diary card
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 35 | 33
Participants | 5 | 2

21. Secondary Outcome: Number of Systemic Events Within 7 Days After Vaccination
Description: Systemic reactions included fever, fatigue, headache, vomiting, nausea, diarrhea, muscle pain, and joint pain. Each of these items was collected on a four-point scale including, none, mild, moderate, and severe.
Time Frame: 7 days post vaccination
Population: The number of participants who completed the vaccination diary card
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 35 | 33
Participants | 18 | 11

22. Secondary Outcome: Number of Participants With an Occurrence of Unsolicited Adverse Events (AEs) Post Vaccination
Description: Number of participants with at least one unsolicited adverse events (AEs) within 30 days after vaccination. Unsolicited AEs were all AEs for which participants were not specifically questioned in the participant diary.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 35 | 35
Participants | 12 | 10

23. Secondary Outcome: Occurrence of Medically Attended AEs
Description: Number of medically attended AEs from vaccination to study end
Time Frame: Through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Groups:
- RSVPreF (From Vaccination Until Viral Challenge): A single intramuscular injection at a dose of 120 mcg reconstituted with sterile water for an 0.5 mL injection volume
  RSVPreF: A single dose of 120 mcg RSVpreF for intramuscular injection on Day -28
- Placebo (From Vaccination Until Viral Challenge): A single intramuscular injection of Placebo to match active vaccine
  Placebo: A single Placebo dose for intramuscular injection to match experimental vaccine on Day -28
- RSVPreF (From Viral Challenge Until Day 28): Participants undergone intranasal challenge with RSV-A Memphis 37b virus on Day 0, after receiving a single intramuscular dose of of 120 mcg RSVpreF on Day -28
- Placebo (From Viral Challenge Until Day 28): Participants undergone intranasal challenge with RSV-A Memphis 37b virus on Day 0, after receiving a single intramuscular dose of placebo on Day -28.
- RSVPreF (From Day 28 Until Day155): Participants completed 6 months post challenge follow up visit after receiving a single intramuscular dose of of 120 mcg RSVpreF on Day -28 and RSV-A Memphis 37b virus on Day 0
- Placebo (From Day 28 Until Day155): Participants completed 6 months post challenge follow up visit after receiving a single intramuscular dose of of Placebo on Day -28 and RSV-A Memphis 37b virus on Day 0
Arm/Group | RSVPreF (From Vaccination Until Viral Challenge) | Placebo (From Vaccination Until Viral Challenge) | RSVPreF (From Viral Challenge Until Day 28) | Placebo (From Viral Challenge Until Day 28) | RSVPreF (From Day 28 Until Day155) | Placebo (From Day 28 Until Day155)
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35 | 35
Participants | 1 | 2 | 2 | 1 | 2 | 0

24. Secondary Outcome: Occurrence of SAEs
Description: Number of SAEs from vaccination to study end
Time Frame: Through study completion, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 35 | 35
Participants | 1 | 1

25. Secondary Outcome: Number of Participants With an Occurrence of Unsolicited AEs Related to Viral Challenge
Description: Number of participants with at least one unsolicited AE within 30 days post-viral challenge (Day 0) up to Day +28 follow up. Unsolicited AEs were all AEs for which participants were not specifically questioned in the participant diary.
Time Frame: Day 0 to Day 28
Population: All vaccinated participants were included in the Safety Analysis Set, irrespective of whether they received challenge virus.
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 35 | 35
Participants | 14 | 17

26. Secondary Outcome: Occurrence of Haematological and Biochemical Laboratory Abnormalities During the Quarantine Period.
Description: Number of hematological and biochemical laboratory assessment Abnormalities reported as AEs during the quarantine period.
Time Frame: Day -2 to Day12
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 35 | 35
Participants
  Mild raised ALT | 8 | 5
  Moderate raised ALT | 1 | 1
  Mild raised AST | 2 | 5
  Moderate raised AST | 1 | 0
  Moderate raised CK | 0 | 1
  Mild low platelets | 0 | 1
  Mild low lymphocytes | 0 | 1
  Moderate low neutrophils | 0 | 1

27. Secondary Outcome: Use of Concomitant Medication
Description: Concomitant medications (prescription and over the counter drugs and supplements that a study participant had taken alongside the study vaccination) were recorded for the period following vaccination (up to viral challenge) and from viral challenge until Day 28..
Time Frame: From Vaccination (Day -28) until Viral Challenge (Day 0), and From Viral Challenge (Day 0) until Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | RSVPreF | Placebo
Number analyzed (Participants) | 35 | 35
Participants
  Concomitant Medications from Vaccination (Day -28) until Viral Challenge (Day 0) | 9 | 11
  Concomitant Medications from Viral Challenge (Day 0) until Day 28 | 14 | 14

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from vaccination (Day -28) up until viral challenge (Day 0 pre-challenge), following viral challenge (Day 0 post-challenge) until Day 28, and from Day 28 until Day 155. Medically attended AEs and SAEs were recorded from vaccination (Day -28) up until viral challenge (Day 0 pre-challenge), following viral challenge (Day 0 post-challenge) until Day 28, and from Day 28 until Day 155.
Arm/Group | RSVPreF (From Vaccination Until Viral Challenge) | Placebo (From Vaccination Until Viral Challenge) | RSVPreF (From Viral Challenge Until Day 28) | Placebo (From Viral Challenge Until Day 28) | RSVPreF (From Day 28 Until Day155) | Placebo (From Day 28 Until Day155)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 0/35 | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35 | 1/35 | 1/35 | 0/35
Other Adverse Events (participants affected / at risk) | 12/35 | 9/35 | 2/35 | 1/35 | 2/35 | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSVPreF (From Vaccination Until Viral Challenge) (N=35) | Placebo (From Vaccination Until Viral Challenge) (N=35) | RSVPreF (From Viral Challenge Until Day 28) (N=35) | Placebo (From Viral Challenge Until Day 28) (N=35) | RSVPreF (From Day 28 Until Day155) (N=35) | Placebo (From Day 28 Until Day155) (N=35)
Myocarditis (Cardiac disorders) | NA | NA | NA | 1 (1) | 0 (0) | NA
Meningitis viral (Infections and infestations) | NA | NA | NA | 0 (0) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSVPreF (From Vaccination Until Viral Challenge) (N=35) | Placebo (From Vaccination Until Viral Challenge) (N=35) | RSVPreF (From Viral Challenge Until Day 28) (N=35) | Placebo (From Viral Challenge Until Day 28) (N=35) | RSVPreF (From Day 28 Until Day155) (N=35) | Placebo (From Day 28 Until Day155) (N=35)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT04785612/Prot_SAP_000.pdf